CLINICAL TRIAL: NCT05048108
Title: Remote Assessment of Cognition, Insulin Resistance and Omega-3 Fatty Acid Biomarkers in Breast Cancer Survivors at Risk for Cognitive Impairment
Brief Title: Remote Assessment of Cognition, Insulin Resistance and Omega-3 Fatty Acid Biomarkers in Breast Cancer Survivors
Acronym: RACIRO-3
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Tonya Orchard, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-21100
Record Dates: First submitted 2021-08-30; First posted 2021-09-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Obesity
Keywords: Chemotherapy; Cognitive impairment; Breast cancer survivor; Diet; Remote assessment
MeSH Terms: conditions — Breast Neoplasms; Obesity; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Majority of breast cancer survivors are overweight or obese at time of diagnosis, putting them at increased risk for insulin resistance and Type 2 Diabetes Mellitus (T2DM). Women with insulin resistance at time of breast cancer diagnosis often have larger tumors, later stages of cancer and worse prognosis. Additionally, chemotherapy often leads to increases in insulin resistance and cognitive impairment. Many cancer survivors experience memory and brain function decline following chemotherapy that can last for years, and insulin resistance may contribute to worse cognitive outcomes in cancer survivors. Omega-3 polyunsaturated fatty acids (PUFAs) are anti-inflammatory nutrients that may help reduce insulin resistance and negative cognitive outcomes from cancer treatments. The purpose of this observational study with cross-sectional design is to investigate the relationship of omega-3 PUFAs with insulin resistance and cognitive function in obese breast cancer survivors. Due to the global pandemic caused by the coronavirus disease of 2019 (COVID-19), this study will be conducted entirely remotely using electronic data collection and remote finger-stick blood sample collection. The study will aim to enroll 80 racially and ethnically diverse female breast cancer survivors (age 45-75) who are postmenopausal, and 1 to 4 years post breast cancer diagnosis. Participants will complete study questionnaires online, and some cognitive tests will be completed through zoom sessions with trained study personnel. Participants will be mailed kits with thorough instructions to complete fingerstick blood sample collections and mail them back to the research lab. Upon receipt of blood samples and completion of all study questionnaires, participation will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer diagnosis
* Between 1-4 years post-breast cancer diagnosis
* Postmenopausal (at least 1 year post-menses)
* Ability to access and use internet resources, including Zoom video calls
* English speaking

Exclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* Unwillingness to complete finger prick for blood collection

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors from the Central Ohio area, including those who were seen at The Ohio State University Wexner Medical Center James Cancer Hospital for cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Determine number of participants with insulin resistance via HOMA-IR from remote dried blood spot collection | One day
  Homeostatic model assessment for insulin resistance (HOMA-IR) is calculated by fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5. Insulin and glucose measures will be obtained from the dried blood spot collection.

SECONDARY OUTCOMES:
Remote assessment of cognition using the Hopkins Verbal Learning Test | One day
  Assess cognition remotely through a zoom session by using the Hopkins Verbal Learning Test (HVLT), a brief cognitive test of episodic memory and verbal learning.
Remote assessment of cognition using the WAIS-IV Digit Span | One day
  Assess cognition remotely through a zoom session by using the Wechsler Adult Intelligence Scale (WAIS)-IV Digit Span, a cognitive test of attention and working memory.
Remote assessment of cognition using the Oral Trail Making Test | One day
  Assess cognition remotely through a zoom session by using the Oral Trail Making Test (TMT), a brief cognitive test of executive function and attention.
Remote assessment of cognition using the COWA Test | One day
  Assess cognition remotely through a zoom session by using the Controlled Oral Word Association (COWA) Test, a brief cognitive test of oral fluency and executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya S Orchard, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu